CLINICAL TRIAL: NCT02700464
Title: The Efficacy of the Bladder EpiCheck for Detection of Recurrent Urothelial Cell Carcinoma: A Multicenter, Prospective Blinded Pivotal Study
Brief Title: The Efficacy of the Bladder EpiCheck for Detection of Recurrent Urothelial Cell Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nucleix Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: UC-EpiCheck-FDA-01
Record Dates: First submitted 2016-02-24; First posted 2016-03-07 (Estimated); Last update posted 2021-05-04 (Actual); Status verified 2020-07

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Cystoscopy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bladder EpiCheck Urine Test (Experimental): Bladder EpiCheck Urine Test
  Interventions: Device: Bladder EpiCheck Urine Test
- Gold Standard (Active Comparator): Cystoscopy and pathology
  Interventions: Procedure: Cystoscopy and pathology

INTERVENTIONS:
Device: Bladder EpiCheck Urine Test — The Bladder EpiCheck test is an in vitro diagnostic device for the detection of DNA methylation patterns in urine that are associated with bladder cancer. It is intended for use as a noninvasive method for monitoring for tumor recurrence in conjunction with cystoscopy inpatients previously diagnosed with bladder cancer
  Arms: Bladder EpiCheck Urine Test
Procedure: Cystoscopy and pathology — Routine cystoscopy for bladder cancer recurrence and pathology confirmation for patients with positive cystoscopy
  Arms: Gold Standard

SUMMARY:
Clinical trial to determine the efficacy (sensitivity and specificity) of the Bladder EpiCheck test compared to the gold standard cystoscopy and pathology in patients under monitoring for recurrence of bladder cancer.

DETAILED DESCRIPTION:
The Bladder EpiCheck test is an in vitro diagnostic device for the detection of DNA methylation patterns in urine that are associated with bladder cancer. It is intended for use as a noninvasive method for monitoring for tumor recurrence in conjunction with cystoscopy inpatients previously diagnosed with bladder cancer This is a, multicenter, prospective, blinded study to evaluate the efficacy (sensitivity and specificity) of a novel methylation test for the detection of recurrent Urothelial Cell Carcinoma in patients with a history of bladder cancer undergoing surveillance.

ELIGIBILITY:
Inclusion Criteria:

* Any male or female patient diagnosed with incident or recurrent Urothelial Cell Carcinoma and undergoing surveillance at 3 month intervals.
* Has had all urothelial cell carcinoma tumor resected within the past 12 months
* Has a plan for cystoscopic surveillance (adjuvant intravesical therapy allowed)
* Able to provide legally effective informed consent
* Able to produce 45mL of urine

Exclusion Criteria:

* Planning to undergo radical cystectomy or chemotherapy-radiation for Urothelial Cell Carcinoma

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 680 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Specificity of Bladder EpiCheck Urine Test Kit (the proportion of negatives that are correctly identified as such by the gold standard) | Day 1
Sensitivity of Bladder EpiCheck Urine Test Kit (The proportion of positives that are correctly identified as such by the gold standard) | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Shmulik Adler, MSc, Study Director — Nucleix Ltd.
Locations (11):
- United States (10):
  - The Urology Center of Colorado, Denver, Colorado
  - Chesapeake Urology Research Associates, Baltimore, Maryland
  - Michigan Institute of Urology, P.C., Troy, Michigan
  - Metro Urology, Woodbury, Minnesota
  - Urological Surgeons of Long Island, Garden City, New York
  - Duke University Health System, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Urology San Antonio, San Antonio, Texas
  - University Of Washington, Seattle, Washington
- UHN, Princess Margret Cancer center, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No